CLINICAL TRIAL: NCT02194699
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Tralokinumab in Adults and Adolescents With Asthma Inadequately Controlled on Inhaled Corticosteroid Plus Long-Acting β2-Agonist
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Tralokinumab in Adults and Adolescents With Uncontrolled Asthma
Acronym: STRATOS2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D2210C00008
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Results first posted 2018-03-21 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Uncontrolled Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tralokinumab (Experimental): Tralokinumab subcutaneous injection
  Interventions: Biological: Experimental: Tralokinumab
- Placebo (Placebo Comparator): Placebo subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Experimental: Tralokinumab — Tralokinumab subcutaneous injection
  Arms: Tralokinumab
Other: Placebo — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
A 52-Week, Multicentre, Randomized, Double-Blind, Parallel Group, Placebo Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Tralokinumab in Adults and Adolescents with Asthma Inadequately Controlled on Inhaled Corticosteroid Plus Long-Acting β2-Agonist

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel group, placebo-controlled study designed to evaluate efficacy and safety of tralokinumab administered subcutaneously in subjects with uncontrolled asthma on inhaled corticosteroid plus long-acting β2-agonist and having a history of asthma exacerbations. Approximately 770 subjects will be randomized globally. Subjects will receive tralokinumab, or placebo, administered via subcutaneous injection at the study site, over a 52-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12 -75
2. Documented physician-diagnosed asthma.
3. Documented treatment with ICS at a total daily dose corresponding to ≥500μg fluticasone propionate dry powder formulation equivalents) and a LABA
4. Morning pre-BD FEV1 value of ≥40 and <80% value (<90% for patients 12 to 17 years of age) of their PNV.
5. Post-BD reversibility of ≥12% and ≥200 mL in FEV1
6. ACQ-6 score ≥1.5

Exclusion Criteria:

1. Pulmonary disease other than asthma
2. History of anaphylaxis following any biologic therapy
3. Hepatitis B, C or HIV
4. Pregnant or breastfeeding
5. History of cancer
6. Current tobacco smoking or a history of tobacco smoking for ≥ 10 pack-years
7. Previous receipt of tralokinumab

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 856 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Brightling, MD, Principal Investigator — Institute for Lung Health, United Kingdom
Locations (199):
- United States (71):
  - Research Site, Birmingham, Alabama
  - Research Site, Hoover, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Bakersfield, California
  - Research Site, Buena Park, California
  - Research Site, Encinitas, California
  - Research Site, Lakewood, California
  - Research Site, Lomita, California
  - Research Site, Northridge, California
  - Research Site, Palmdale, California
  - Research Site, Roseville, California
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, Thousand Oaks, California
  - Research Site, Ventura, California
  - Research Site, Walnut Creek, California
  - Research Site, Centennial, Colorado
  - Research Site, Celebration, Florida
  - Research Site, DeLand, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palmetto Bay, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Eagle, Idaho
  - Research Site, Evergreen Park, Illinois
  - Research Site, Kenilworth, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, White Marsh, Maryland
  - Research Site, Fall River, Massachusetts
  - Research Site, Reno, Nevada
  - Research Site, Northfield, New Jersey
  - Research Site, Ocean City, New Jersey
  - Research Site, Teaneck, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Verona, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Larchmont, New York
  - Research Site, The Bronx, New York
  - Research Site, Wappingers Falls, New York
  - Research Site, Burlington, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Rock Hill, South Carolina
  - Research Site, Arlington, Texas
  - Research Site, Baytown, Texas
  - Research Site, Frisco, Texas
  - Research Site, Houston, Texas
  - Research Site, Kingwood, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Orem, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Fairfax, Virginia
  - Research Site, Greenfield, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Canada (13):
  - Research Site, Sherwood Park, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Chile (2):
  - Research Site, Santiago
  - Research Site, Talcahuano
- Czechia (6):
  - Research Site, Brandýs nad Labem
  - Research Site, Jindřichův Hradec
  - Research Site, Prague
  - Research Site, Praha 10 - Strasnice
  - Research Site, Rokycany
  - Research Site, Teplice
- Italy (10):
  - Research Site, Catania
  - Research Site, Genova
  - Research Site, Legnago
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Pisa
  - Research Site, Salerno
  - Research Site, Verona
- Japan (42):
  - Research Site, Asahi-shi
  - Research Site, Chūōku
  - Research Site, Fukui-shi
  - Research Site, Fukushima
  - Research Site, Habikino-shi
  - Research Site, Himeji-shi
  - Research Site, Hiroshima
  - Research Site, Itabashi-ku
  - Research Site, Izumo-shi
  - Research Site, Kagoshima
  - Research Site, Kanazawa
  - Research Site, Kanuma-shi
  - Research Site, Kasuga-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kobe
  - Research Site, Kochi
  - Research Site, Maebashi
  - Research Site, Matsue
  - Research Site, Matsusaka-shi
  - Research Site, Meguro-ku
  - Research Site, Minatoku
  - Research Site, Morioka
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Nishinomiya-shi
  - Research Site, Sagamihara-shi
  - Research Site, Sakaide-shi
  - Research Site, Sapporo
  - Research Site, Sasebo-shi
  - Research Site, Seto-shi
  - Research Site, Shibuya-ku
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Sumida-ku
  - Research Site, Takamatsu
  - Research Site, Toshima-ku
  - Research Site, Touon-shi
  - Research Site, Toyama
  - Research Site, Tsu
  - Research Site, Tsukubo-gun
  - Research Site, Uozu-shi
  - Research Site, Yokohama
- Mexico (4):
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Villahermosa
- Philippines (6):
  - Research Site, Caloocan
  - Research Site, Iloilo City
  - Research Site, Lipa City
  - Research Site, Pasig
  - Research Site, Quezon City
  - Research Site, San Fernando City
- Russia (15):
  - Research Site, Chelyabinsk
  - Research Site, Izhevsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Perm
  - Research Site, Petrozavodsk
  - Research Site, Pyatigorsk
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Ulyanovsk
  - Research Site, Vladikavkaz
  - Research Site, Volgograd
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- South Africa (6):
  - Research Site, Boksburg North
  - Research Site, Durban
  - Research Site, KwaDukuza
  - Research Site, Mount Edgecombe
  - Research Site, Mowbray
  - Research Site, Port Elizabeth
- Taiwan (3):
  - Research Site, Kaohsiung Hsien
  - Research Site, Keelung
  - Research Site, New Taipei City
- Ukraine (11):
  - Research Site, Cherkasy
  - Research Site, Dnipropetrovsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kremenchuk
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Sumy
  - Research Site, Uzhhorod
  - Research Site, Zaporizhzhya
- United Kingdom (10):
  - Research Site, Bradford
  - Research Site, Cambridge
  - Research Site, Chertsey
  - Research Site, Glasgow
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, Manchester
  - Research Site, Northwood
  - Research Site, Sidcup
  - Research Site, Wishaw

IPD SHARING:
Plan to Share IPD: No
This is commercially sensitive information.

REFERENCES:
- [Derived] Gottlow M, Svensson DJ, Lipkovich I, Huhn M, Bowen K, Wessman P, Colice G. Application of structured statistical analyses to identify a biomarker predictive of enhanced tralokinumab efficacy in phase III clinical trials for severe, uncontrolled asthma. BMC Pulm Med. 2019 Jul 17;19(1):129. doi: 10.1186/s12890-019-0889-4. PMID 31315668
- [Derived] Carlsson M, Braddock M, Li Y, Wang J, Xu W, White N, Megally A, Hunter G, Colice G. Evaluation of Antibody Properties and Clinically Relevant Immunogenicity, Anaphylaxis, and Hypersensitivity Reactions in Two Phase III Trials of Tralokinumab in Severe, Uncontrolled Asthma. Drug Saf. 2019 Jun;42(6):769-784. doi: 10.1007/s40264-018-00788-w. PMID 30649752
- [Derived] Panettieri RA Jr, Sjobring U, Peterffy A, Wessman P, Bowen K, Piper E, Colice G, Brightling CE. Tralokinumab for severe, uncontrolled asthma (STRATOS 1 and STRATOS 2): two randomised, double-blind, placebo-controlled, phase 3 clinical trials. Lancet Respir Med. 2018 Jul;6(7):511-525. doi: 10.1016/S2213-2600(18)30184-X. Epub 2018 May 20. PMID 29792288
- [Derived] Panettieri RA Jr, Wang M, Braddock M, Bowen K, Colice G. Tralokinumab for the treatment of severe, uncontrolled asthma: the ATMOSPHERE clinical development program. Immunotherapy. 2018 Mar 1;10(6):473-490. doi: 10.2217/imt-2017-0191. Epub 2018 Mar 14. PMID 29536781

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 30 Oct 2014; Last Patient Last Visit: 21 Sep 2017. Study performed at 242 sites in 13 countries.
  Patients were maintained on their currently prescribed inhaled corticosteroid long-acting β2-agonist therapy and any additional maintenance asthma controller medications throughout the study period.
Pre-assignment Details: 1696 patients signed informed consent, 1163 entered screening/run-in period, 856 patients were randomised to receive investigational product (IP) and 849 received treatment.
  The primary population was the biomarker positive population, defined as all patients with baseline fractional exhaled nitric oxide (FeNO) ≥37 parts per billion (ppb).
Groups:
- Tralo 300 mg Q2W: Tralokinumab 300 milligrams (mg) administered subcutaneously every 2 weeks (Q2W) over a 52-week treatment period (up to 26 doses).
- Placebo: Placebo administered subcutaneously Q2W over a 52-week treatment period (up to 26 doses).
Period: Randomised
Arm/Group | Tralo 300 mg Q2W | Placebo
Started | 428 | 428
Completed | 420 | 417
Not Completed | 8 | 11
Not completed — Did not receive treatment | 1 | 5
Not completed — Without potential for 52 weeks of IP | 5 | 5
Not completed — Duplicate patient | 2 | 1
Period: With Potential to Receive 52 Weeks of IP
Arm/Group | Tralo 300 mg Q2W | Placebo
Started | 420 (Includes all patients randomised with the potential to receive 52 weeks of IP and receiving any IP.) | 417 (Includes all patients randomised with the potential to receive 52 weeks of IP and receiving any IP.)
Completed | 370 | 365
Not Completed | 50 | 52
Not completed — Adverse Event | 4 | 3
Not completed — Death | 1 | 3
Not completed — Lost to Follow-up | 5 | 8
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 14 | 20
Not completed — Other | 24 | 16

BASELINE CHARACTERISTICS:
Population: All patients in the full analysis set (FAS) with the potential to receive 52 weeks of IP and who received any IP (tralokinumab or placebo) were included in the baseline analysis.
Groups:
- Tralo 300 mg Q2W: Tralokinumab 300 mg administered subcutaneously Q2W over a 52-week treatment period (up to 26 doses).
- Total: Total of all reporting groups
Arm/Group | Tralo 300 mg Q2W | Placebo | Total
Number analyzed (Participants) | 420 | 417 | 837
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.3 (15.6) | 48.0 (15.5) | 47.6 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 276 | 290 | 566
  Male | 144 | 127 | 271
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 83 | 88 | 171
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 24 | 51
  White | 283 | 281 | 564
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 24 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: Annualised Asthma Exacerbation Rate (AAER) up to Week 52
Description: Asthma exacerbation was defined as a worsening of asthma that led to any of the following:
  * Use of systemic corticosteroids for at least 3 days; a single depo-injectable dose of corticosteroids was considered equivalent to a 3-day course of systemic corticosteroids.
  * An emergency room (ER) or urgent care (UC) visit (defined as evaluation and treatment for <24 hours in an ER or UC centre) due to asthma that required systemic corticosteroids (see above).
  * An inpatient hospitalisation (defined as admission to an inpatient facility and/or evaluation and treatment in a healthcare facility for ≥24 hours) due to asthma.
  AAER = number of exacerbations*365.25 / (follow-up date - date of randomisation + 1) (where maximum follow-up time for a patient was approximately 52 weeks).
  AAER in the tralokinumab group was compared to that seen in the placebo group up to Week 52 using a negative binomial model; rate ratios and rate reductions are both presented for comparative statistical analyses.
Time Frame: Baseline (Week 0) up to Week 52
Population: The FAS included all randomised patients with the potential to receive 52 weeks of IP and receiving any IP, irrespective of their protocol adherence and continued participation in the study.
Measure: Number (95% Confidence Interval); unit: Events/year
Groups:
- Biomarker Positive - Tralo 300 mg Q2W: Tralokinumab 300 mg administered subcutaneously Q2W over a 52-week treatment period (up to 26 doses). Patients in the biomarker positive population (primary population) had baseline FeNO ≥37 ppb.
- Biomarker Positive - Placebo: Placebo administered subcutaneously Q2W over a 52-week treatment period (up to 26 doses). Patients in the biomarker positive population (primary population) had baseline FeNO ≥37 ppb.
- Biomarker Negative - Tralo 300 mg Q2W: Tralokinumab 300 mg administered subcutaneously Q2W over a 52-week treatment period (up to 26 doses). Patients in the biomarker negative population (complement population) had baseline FeNO <37 ppb.
- Biomarker Negative - Placebo: Placebo administered subcutaneously Q2W over a 52-week treatment period (up to 26 doses). Patients in the biomarker negative population (complement population) had baseline FeNO <37 ppb.
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 108 | 121 | 308 | 290 | 420 | 417
Events/year | 0.80 [0.57 to 1.11] | 0.95 [0.68 to 1.31] | 0.87 [0.71 to 1.06] | 0.77 [0.63 to 0.95] | 0.84 [0.71 to 1.00] | 0.82 [0.69 to 0.97]
Statistical Analysis 1: Comparison: Biomarker Positive - Tralo 300 mg Q2W vs Biomarker Positive - Placebo; Comparison of AAER (rate ratio): Biomarker positive population; Tralo 300 mg Q2W vs placebo. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term was included in the analysis model; Test type: Superiority — The null hypothesis was that the exacerbation rate during the 52-week double-blind treatment period on tralokinumab was equal to the corresponding exacerbation rate on placebo; p = 0.4656, Negative binomial; Rate ratio = 0.84, 95% CI 2-sided [0.53 to 1.34] — Covariates in the model included treatment group, geographical region, age group, periostin group at baseline and number of exacerbations in the year before the study
Statistical Analysis 2: Comparison: Biomarker Negative - Tralo 300 mg Q2W vs Biomarker Negative - Placebo; Comparison of AAER (rate ratio): Biomarker negative population; Tralo 300 mg Q2W vs placebo. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term was included in the analysis model; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4126, Negative binomial; Rate ratio = 1.13, 95% CI 2-sided [0.85 to 1.50] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Biomarker Positive - Tralo 300 mg Q2W vs Biomarker Positive - Placebo; Comparison of AAER (rate reduction): Biomarker positive population; Tralo 300 mg Q2W vs placebo. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term was included in the analysis model; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4656, Negative binominal; Rate reduction = 15.83, 95% CI 2-sided [-33.71 to 47.01] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of AAER (rate ratio): FAS population; Tralo 300 mg Q2W vs placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8027, Negative binomial; Rate ratio = 1.03, 95% CI 2-sided [0.81 to 1.31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of AAER (rate reduction): FAS population; Tralo 300 mg Q2W vs placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8027, Negative binominal; Rate reduction = -3.14, 95% CI 2-sided [-31.46 to 19.08] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percent Change From Baseline to Week 52 in Pre-dose/Pre-bronchodilator (BD) Forced Expiratory Volume in 1 Second (FEV1)
Description: Lung function was assessed by FEV1 which was measured by spirometry. Spirometry was performed by the Investigator or authorised delegate according to American Thoracic Society/European Respiratory Society guidelines. The mean percent change from baseline in pre-BD FEV1 at Week 52 is presented.
Time Frame: Baseline (Week 0) and Week 52
Population: The FAS included all randomised patients with the potential to receive 52 weeks of IP and receiving any IP, irrespective of their protocol adherence and continued participation in the study. Only patients with data available at the timepoints of testing were included in the analyses.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 99 | 103 | 282 | 250 | 384 | 358
Percent change from baseline | 18.769 (29.628) | 16.632 (31.906) | 13.103 (24.641) | 8.395 (21.962) | 14.546 (26.065) | 10.528 (25.475)
Statistical Analysis 1: Comparison: Biomarker Positive - Tralo 300 mg Q2W vs Biomarker Positive - Placebo; Comparison of % change from baseline in pre-dose/pre-BD FEV1 at Week 52: Biomarker positive population; Tralo 300 mg Q2W vs placebo. Restricted maximum likelihood (REML) based repeated measures analysis on patients with a baseline pre-dose/pre-BD FEV1 assessment. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.6033, Repeated measures analysis; Least square (LS) Mean difference = 1.86, 95% CI 2-sided [-5.16 to 8.88] — Fixed categorical effects of treatment group, geographical region, age group, periostin group, visit and treatment-by-visit interaction and number of asthma exacerbations in year before study as a fixed covariate
Statistical Analysis 2: Comparison: Biomarker Negative - Tralo 300 mg Q2W vs Biomarker Negative - Placebo; Comparison of % change from baseline in pre-dose/pre-BD FEV1 at Week 52: Biomarker negative population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis on patients with a baseline pre-dose/pre-BD FEV1 assessment. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.1276, Repeated measures analysis; LS Mean difference = 3.37, 95% CI 2-sided [-0.97 to 7.70] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of % change from baseline in pre-dose/pre-BD FEV1 at Week 52: FAS population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis on patients with a baseline pre-dose/pre-BD FEV1 assessment; Test type: Superiority; p = 0.1164, Repeated measures analysis; LS Mean difference = 2.95, 95% CI 2-sided [-0.73 to 6.62] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Change From Baseline to Week 52 in Total Asthma Symptom Score (Bi-weekly Means)
Description: Asthma symptoms during night-time and daytime were recorded by the patient each morning and evening in the Asthma Daily Diary. Symptoms were recorded using a 4-point response scale, which ranged from 0 to 3, where 0 indicated no asthma symptoms. Asthma symptom daytime score (recorded in the evening), night-time score (recorded in the morning), and total score were calculated separately. The daily asthma symptom total score was calculated by taking the sum of the night-time and daytime asthma symptom scores recorded each day, ranging from 0 to 6. A lower symptom score indicated a better outcome. The change from baseline in bi-weekly mean daily asthma symptom total score is presented.
Time Frame: Baseline (Week 0) and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 79 | 81 | 215 | 223 | 297 | 309
Scores on a scale | -1.18 (0.98) | -1.06 (1.25) | -0.98 (1.04) | -1.02 (1.24) | -1.04 (1.04) | -1.02 (1.24)
Statistical Analysis 1: Comparison: Biomarker Positive - Tralo 300 mg Q2W vs Biomarker Positive - Placebo; Comparison of mean change from baseline in total asthma symptom score at Week 52: Biomarker positive population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.1456, Repeated measures analysis; LS Mean difference = -0.20, 95% CI 2-sided [-0.47 to 0.07] — Fixed categorical effects of baseline asthma symptom score, treatment group, geographical region, age group, periostin group, visit and treatment-by-visit interaction and number of asthma exacerbations in year before study as a fixed covariate
Statistical Analysis 2: Comparison: Biomarker Negative - Tralo 300 mg Q2W vs Biomarker Negative - Placebo; Comparison of mean change from baseline in total asthma symptom score at Week 52: Biomarker negative population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.6548, Repeated measures analysis; LS Mean difference = 0.04, 95% CI 2-sided [-0.13 to 0.20] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of mean change from baseline in total asthma symptom score at Week 52: FAS population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis; Test type: Superiority; p = 0.5763, Repeated measures analysis; LS Mean difference = -0.04, 95% CI 2-sided [-0.18 to 0.10] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline to Week 52 in Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ(S)+12) Total Score
Description: The AQLQ(S)+12 is a questionnaire that measures health-related quality of life for patients with asthma aged 12 and older. The questionnaire comprises 32 questions and has 4 separate domains (asthma symptoms, activity limitations, emotional function and environmental stimuli). Patients were asked to recall their experiences during the previous 2 weeks and to score each of the questions on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment). The total score was calculated as the mean response to all questions, ranging from 1 (severe impairment) to 7 (no impairment). Individual AQLQ(S)+12 total score changes of ≥0.5 were considered to be clinically meaningful. The mean change from baseline in AQLQ(S)+12 score at Week 52 is presented.
Time Frame: Baseline (Week 0) and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 77 | 84 | 242 | 230 | 321 | 318
Scores on a scale | 1.35 (1.06) | 1.20 (1.22) | 1.13 (1.07) | 1.23 (1.25) | 1.18 (1.07) | 1.21 (1.24)
Statistical Analysis 1: Comparison: Biomarker Positive - Tralo 300 mg Q2W vs Biomarker Positive - Placebo; Comparison of change in mean score from baseline for AQLQ(S)+12 at Week 52: Biomarker positive population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.0874, Repeated measures analysis; LS Mean difference = 0.27, 95% CI 2-sided [-0.04 to 0.57] — Fixed categorical effects of baseline AQLQ(S)+12 score, treatment group, geographical region, age group, periostin group, visit and treatment-by-visit interaction and number of asthma exacerbations in year before study as a fixed covariate
Statistical Analysis 2: Comparison: Biomarker Negative - Tralo 300 mg Q2W vs Biomarker Negative - Placebo; Comparison of change in mean score from baseline for AQLQ(S)+12 at Week 52: Biomarker negative population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.9083, Repeated measures analysis; LS Mean difference = -0.01, 95% CI 2-sided [-0.20 to 0.17] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of change in mean score from baseline for AQLQ(S)+12 at Week 52: FAS population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis; Test type: Superiority; p = 0.4506, Repeated measures analysis; LS Mean difference = 0.06, 95% CI 2-sided [-0.10 to 0.22] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline to Week 52 in Asthma Control Questionnaire-6 (ACQ-6) Score
Description: The ACQ-6 questionnaire is a shortened version of the ACQ (omitting FEV1 measurement) that assesses asthma symptoms (night-time awakenings, symptoms on waking, activity limitation, dyspnoea, wheezing) and rescue short-acting β2-agonists medication use during the past week. Questions were weighted equally and scored on a 7-point scale from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-6 score was the mean of the responses, ranging from 0 (totally controlled) to 6 (severely uncontrolled). Mean scores of ≤0.75 indicate well-controlled asthma, scores between 0.75 and ≤1.5 indicate partly controlled asthma and a score >1.5 indicates not well-controlled asthma. Individual changes of at least 0.5 were considered to be clinically meaningful. The mean change from baseline in ACQ-6 score at Week 52 is presented.
Time Frame: Baseline (Week 0) and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 85 | 86 | 254 | 243 | 341 | 334
Scores on a scale | -1.26 (1.01) | -1.14 (1.12) | -1.07 (1.02) | -1.11 (1.13) | -1.12 (1.02) | -1.11 (1.13)
Statistical Analysis 1: Comparison: Biomarker Positive - Tralo 300 mg Q2W vs Biomarker Positive - Placebo; Comparison of change in mean score from baseline for ACQ-6 at Week 52: Biomarker positive population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.0400, Repeated measures analysis; LS Mean difference = -0.27, 95% CI 2-sided [-0.53 to -0.01] — Fixed categorical effects of baseline ACQ-6 score, treatment group, geographical region, age group, periostin group, visit and treatment-by-visit interaction and number of asthma exacerbations in year before study as a fixed covariate
Statistical Analysis 2: Comparison: Biomarker Negative - Tralo 300 mg Q2W vs Biomarker Negative - Placebo; Comparison of change in mean score from baseline for ACQ-6 at Week 52: Biomarker negative population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.9735, Repeated measures analysis; LS Mean difference = 0.00, 95% CI 2-sided [-0.16 to 0.16] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of change in mean score from baseline for ACQ-6 at Week 52: FAS population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis; Test type: Superiority; p = 0.2432, Repeated measures analysis; LS Mean difference = -0.08, 95% CI 2-sided [-0.21 to 0.05] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: AAER Associated With an ER/UC Visit, or a Hospitalisation up to Week 52
Description: The annual rate of exacerbations associated with an ER/UC visit or hospitalisation up to Week 52 are presented for non-adjudicated data (i.e. events assessed by the Investigator and recorded in the electronic case report form).
  AAER = number of exacerbations*365.25 / (follow-up date - date of randomisation + 1) (where maximum follow-up time for a patient was approximately 52 weeks).
Time Frame: Baseline (Week 0) up to Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events/year
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 108 | 121 | 308 | 290 | 420 | 417
Events/year | 0.06 [0.03 to 0.14] | 0.16 [0.09 to 0.29] | 0.09 [0.06 to 0.14] | 0.11 [0.07 to 0.17] | 0.08 [0.06 to 0.12] | 0.12 [0.09 to 0.18]
Statistical Analysis 1: Comparison: Biomarker Positive - Tralo 300 mg Q2W vs Biomarker Positive - Placebo; Comparison of AAER associated with an ER/UC visit or hospitalisation: Biomarker positive population; Tralo 300 mg Q2W vs placebo. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term was included in the analysis model; Test type: Superiority; p = 0.0576, Negative binomial; Rate ratio = 0.39, 95% CI 2-sided [0.15 to 1.03] — Covariates in the model included treatment group, geographical region, age group, periostin group at baseline and number of exacerbations resulting in hospitalisation or ER treatment (yes/no) in the year before the study
Statistical Analysis 2: Comparison: Biomarker Negative - Tralo 300 mg Q2W vs Biomarker Negative - Placebo; Comparison of AAER associated with an ER/UC visit or hospitalisation: Biomarker negative population; Tralo 300 mg Q2W vs placebo. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term was included in the analysis model; Test type: Superiority; p = 0.5249, Negative binomial; Rate ratio = 0.83, 95% CI 2-sided [0.46 to 1.48] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of AAER associated with an ER/UC visit or hospitalisation: FAS population; Tralo 300 mg Q2W vs placebo; Test type: Superiority; p = 0.1155, Negative binomial; Rate ratio = 0.67, 95% CI 2-sided [0.41 to 1.10] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Change From Baseline in European Quality of Life - 5 Dimension 5 Levels (EQ-5D-5L) Visual Analogue Scale (VAS) Scores at Week 52
Description: The EQ-5D-5L questionnaire assesses 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response options (no problems, slight problems, moderate problems, severe problems and extreme problems) that reflect increasing levels of difficulty. The patient was asked to indicate his/her current health state by selecting the most appropriate level in each of the 5 dimensions. The questionnaire also included a VAS, where the patient was asked to rate current health status on a scale of 0 to 100, with 0 being the worst imaginable health state. The mean change from baseline in EQ-5D-5L VAS scores at Week 52 is presented.
Time Frame: Baseline (Week 0) and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 81 | 85 | 233 | 224 | 317 | 313
Scores on a scale | 14.58 (15.21) | 11.58 (17.26) | 11.67 (17.18) | 12.01 (17.43) | 12.46 (16.67) | 11.66 (17.41)

8. Secondary Outcome: Change From Baseline in Total Asthma Rescue Medication Use at Week 52 (Bi-weekly Means)
Description: Salbutamol, albuterol or levalbuterol were used as rescue medication during the study in the event of a worsening of asthma symptoms. Rescue medication use was measured by the bi-weekly mean number of inhalations (puffs) per day, calculated as: total morning puffs + total evening puffs + 2*(total morning nebuliser use + total evening nebuliser use)/ total number of days with data in bi-weekly period. The change from baseline in bi-weekly mean total asthma rescue medication use at Week 52 is presented.
Time Frame: Baseline (Week 0) and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Puffs/day
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 79 | 81 | 215 | 223 | 297 | 309
Puffs/day | -2.86 (3.26) | -1.73 (4.59) | -2.01 (2.93) | -2.08 (4.28) | -2.25 (3.03) | -1.97 (4.34)
Statistical Analysis 1: Comparison: Biomarker Positive - Tralo 300 mg Q2W vs Biomarker Positive - Placebo; Comparison of mean change from baseline in rescue medication use at Week 52: Biomarker positive population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.0360, Repeated measures analysis; LS Mean difference = -0.95, 95% CI 2-sided [-1.85 to -0.06] — Fixed categorical effects of baseline rescue medication use, treatment group, geographical region, age group, periostin group, visit and treatment-by-visit interaction and number of asthma exacerbations in year before study as a fixed covariate
Statistical Analysis 2: Comparison: Biomarker Negative - Tralo 300 mg Q2W vs Biomarker Negative - Placebo; Comparison of mean change from baseline in rescue medication use at Week 52: Biomarker negative population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.5864, Repeated measures analysis; LS Mean difference = 0.15, 95% CI 2-sided [-0.40 to 0.70] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of mean change from baseline in rescue medication use at Week 52: FAS population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis; Test type: Superiority; p = 0.4689, Repeated measures analysis; LS Mean difference = -0.17, 95% CI 2-sided [-0.63 to 0.29] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Change From Baseline in Home Peak Expiratory Flow (PEF) (Morning and Evening) at Week 52
Description: Home PEF testing was performed by the patient using an electronic, hand-held spirometer (peak flow meter) and was performed in the morning upon awakening (prior to taking their morning asthma controller) and in the evening at bedtime (prior to taking their evening asthma controller). The mean change from baseline in home PEF values at Week 52 are presented separately for morning and evening.
Time Frame: Baseline (Week 0) and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 86 | 86 | 233 | 222 | 322 | 313
L/min
  Morning PEF: number analyzed (Participants) | 84 | 81 | 231 | 222 | 318 | 308
  Morning PEF | 22.35 (74.00) | 18.80 (86.24) | 6.72 (73.82) | 6.10 (72.28) | 10.66 (73.88) | 9.43 (76.01)
  Evening PEF | 18.15 (69.20) | 8.88 (79.72) | 1.72 (79.58) | 0.17 (73.66) | 5.72 (77.01) | 2.91 (74.94)
Statistical Analysis 1: Comparison: Biomarker Positive - Tralo 300 mg Q2W vs Biomarker Positive - Placebo; Comparison of mean change from baseline in morning PEF at Week 52: Biomarker positive population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.5094, Repeated measures analysis; LS Mean difference = 6.15, 95% CI 2-sided [-12.13 to 24.43] — Fixed categorical effects of baseline PEF (morning), treatment group, geographical region, age group, periostin group, visit and treatment-by-visit interaction and number of asthma exacerbations in year before study as a fixed covariate
Statistical Analysis 2: Comparison: Biomarker Negative - Tralo 300 mg Q2W vs Biomarker Negative - Placebo; Comparison of mean change from baseline in morning PEF at Week 52: Biomarker negative population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.5984, Repeated measures analysis; LS Mean difference = 3.02, 95% CI 2-sided [-8.22 to 14.26] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Biomarker Positive - Tralo 300 mg Q2W vs Biomarker Positive - Placebo; Comparison of mean change from baseline in evening PEF at Week 52: Biomarker positive population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.3971, Repeated measures analysis; LS Mean difference = 7.84, 95% CI 2-sided [-10.32 to 26.00] — Model included fixed categorical effects of baseline PEF (evening), treatment group, geographical region, age group, periostin group, visit and treatment-by-visit interaction and number of asthma exacerbations in year before study as fixed covariate
Statistical Analysis 4: Comparison: Biomarker Negative - Tralo 300 mg Q2W vs Biomarker Negative - Placebo; Comparison of mean change from baseline in evening PEF at Week 52: Biomarker negative population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.5310, Repeated measures analysis; LS Mean difference = 3.59, 95% CI 2-sided [-7.65 to 14.83] — [estimate comment as in outcome 9, analysis 3]
Statistical Analysis 5: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of mean change from baseline in morning PEF at Week 52: FAS population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis; Test type: Superiority; p = 0.4764, Repeated measures analysis; LS Mean difference = 3.46, 95% CI 2-sided [-6.06 to 12.97] — Model included fixed categorical effects of baseline PEF (morning), treatment group, geographical region, age group, periostin group, visit and treatment-by-visit interaction and number of asthma exacerbations in year before study as fixed covariate
Statistical Analysis 6: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of mean change from baseline in evening PEF at Week 52: FAS population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis; Test type: Superiority; p = 0.4221, Repeated measures analysis; LS Mean difference = 3.88, 95% CI 2-sided [-5.60 to 13.37] — [estimate comment as in outcome 9, analysis 3]

10. Secondary Outcome: Change From Baseline in Night-time Awakenings Due to Asthma Requiring Rescue Medication Use at Week 52 (Bi-weekly Means [Percentage])
Description: The patient captured night-time awakenings (yes/no) and the use of rescue medication during these awakenings (yes/no) each morning in the Asthma Daily Diary. Night-time awakenings (percentage) was defined as the number of nights with awakenings due to asthma and requiring rescue medication divided by number of nights with data. The change from baseline in bi-weekly means (percentage) night-time awakenings due to asthma requiring rescue medication use at Week 52 is presented.
Time Frame: Baseline (Week 0) and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of nights with awakenings
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 94 | 96 | 270 | 247 | 368 | 348
Percentage of nights with awakenings | -37.86 (38.36) | -34.06 (34.96) | -34.65 (34.34) | -35.67 (37.37) | -35.60 (35.40) | -35.05 (36.63)
Statistical Analysis 1: Comparison: Biomarker Positive - Tralo 300 mg Q2W vs Biomarker Positive - Placebo; Comparison of mean change from baseline in number (%) of awakenings at Week 52: Biomarker positive population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis. A variable for the biomarker population (positive, negative) as well as a treatment-by-biomarker population interaction term and a 3-way biomarker population-by-treatment-by-visit interaction term was included in the analysis model; Test type: Superiority; p = 0.1099, Repeated measures analysis; LS Mean difference = -5.04, 95% CI 2-sided [-11.21 to 1.14] — Fixed categorical effects of baseline number (%) of awakenings, treatment group, geographical region, age group, periostin group, visit and treatment-by-visit interaction and number of asthma exacerbations in year before study as a fixed covariate
Statistical Analysis 2: Comparison: Biomarker Negative - Tralo 300 mg Q2W vs Biomarker Negative - Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.8112, Repeated measures analysis; LS Mean difference = 0.46, 95% CI 2-sided [-3.33 to 4.25] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of mean change from baseline in number (%) of awakenings at Week 52: FAS population; Tralo 300 mg Q2W vs placebo. REML based repeated measures analysis; Test type: Superiority; p = 0.4645, Repeated measures analysis; LS Mean difference = -1.19, 95% CI 2-sided [-4.40 to 2.01] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Number of Patients With ≥1 Asthma Exacerbation up to Week 52
Description: The number of patients with ≥1 asthma exacerbation up to Week 52 is presented.
Time Frame: Baseline (Week 0) up to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 108 | 121 | 308 | 290 | 420 | 417
Participants | 38 | 50 | 125 | 117 | 163 | 171
Statistical Analysis 1: Comparison: Biomarker Positive - Tralo 300 mg Q2W vs Biomarker Positive - Placebo; Comparison of number of patients with ≥ 1 asthma exacerbations up to Week 52: Biomarker positive population; Tralo 300 mg Q2W vs placebo; Test type: Superiority; p = 0.3440, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.44 to 1.33] — The estimate of each odds ratio was obtained from a Cochran-Mantel-Haenszel test controlling for geographical region, age group and periostin group at baseline
Statistical Analysis 2: Comparison: Biomarker Negative - Tralo 300 mg Q2W vs Biomarker Negative - Placebo; Comparison of number of patients with ≥ 1 asthma exacerbations up to Week 52: Biomarker negative population; Tralo 300 mg Q2W vs placebo; Test type: Superiority; p = 0.7768, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.75 to 1.46] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of number of patients with ≥ 1 asthma exacerbations up to Week 52: FAS population; Tralo 300 mg Q2W vs placebo; Test type: Superiority; p = 0.5276, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.69 to 1.21] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire and Classroom Impairment Questions (WPAI+CIQ): Productivity Loss at Week 52
Description: The WPAI+CIQ consists of questions about how asthma and asthma-related issues impact a patient's ability to work, attend classes and perform regular daily activities. The questionnaire contains 10 questions relating to the patient's experience over the previous 7 days.
  The WPAI+CIQ outcomes for productivity loss are presented separately for those currently employed and for those currently in school and are expressed as mean productivity loss (percentage) at Week 52, with higher numbers indicating less productivity.
  Work Productivity Loss = {Q2/(Q2+Q4)+[(1-Q2/(Q2+Q4))x(Q5/10)]}*100 (Absenteeism = Q2/(Q2+Q4)*100; Presenteeism = (Q5/10)*100).
  Class Productivity Loss = {Q7/(Q7+Q8) + [(1-Q7/(Q7+Q8))x(Q9/10)]}*100 (Absenteeism = Q7/(Q7+Q8)*100; Presenteeism = (Q9/10)*100).
  Note: QX refers to response to question number X on WPAI+CIQ questionnaire.
Time Frame: At Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent productivity loss
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 46 | 46 | 105 | 104 | 154 | 151
Percent productivity loss
  Productivity loss - currently employed: number analyzed (Participants) | 43 | 34 | 92 | 90 | 137 | 125
  Productivity loss - currently employed | 22.51 (24.47) | 28.15 (27.39) | 23.36 (23.39) | 31.05 (27.20) | 23.43 (23.66) | 30.17 (27.08)
  Productivity loss - currently in school: number analyzed (Participants) | 3 | 12 | 13 | 14 | 17 | 26
  Productivity loss - currently in school | 28.89 (34.21) | 37.92 (28.72) | 25.99 (32.17) | 19.67 (29.06) | 28.03 (31.01) | 28.09 (29.80)

13. Secondary Outcome: WPAI+CIQ: Activity Impairment at Week 52
Description: The WPAI+CIQ consists of questions about how asthma and asthma-related issues impact a patient's ability to work, attend classes and perform regular daily activities. The questionnaire contains 10 questions relating to the patient's experience over the previous 7 days.
  The WPAI+CIQ outcomes for activity impairment are presented separately for those currently employed and for those currently in school and are expressed as mean impairment percentages at Week 52, with higher numbers indicating greater impairment.
  Activity impairment = (Q10/10)*100. Note: QX refers to response to question number X on WPAI+CIQ questionnaire.
Time Frame: At Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent impairment
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 50 | 49 | 116 | 110 | 169 | 160
Percent impairment
  Activity Impairment - currently employed: number analyzed (Participants) | 45 | 36 | 100 | 94 | 147 | 131
  Activity Impairment - currently employed | 20.89 (18.81) | 25.28 (28.63) | 20.50 (20.42) | 26.49 (23.59) | 20.68 (19.82) | 26.11 (24.89)
  Activity Impairment - currently in school: number analyzed (Participants) | 5 | 13 | 16 | 16 | 22 | 29
  Activity Impairment - currently in school | 20.00 (18.71) | 33.85 (26.63) | 26.88 (30.49) | 23.13 (30.27) | 24.55 (27.38) | 27.93 (28.71)

14. Secondary Outcome: Asthma-related Healthcare Encounters by Type up to Week 52
Description: Broad-based healthcare utilisation asthma-related event information was collected by the Investigator/authorised delegate at each visit. At Visit 1, healthcare resource utilisation information was collected with a 1-year recall period; subsequent visits collected information with a recall period of 'since the last scheduled visit'. Total number of times the healthcare encounter occurred was calculated across all patients for each of the following categories:
  * Ambulance transport,
  * Emergency room visits,
  * Unscheduled outpatient visits (visit to specialist and/or visit to primary healthcare physician and/or other healthcare visit),
  * Home visits (home visit, physician and/or other healthcare professional),
  * Telephone calls (telephone calls to physician and/or nurse), and
  * Advanced pulmonary function test.
Time Frame: Baseline (Week 0) up to Week 52
Population: as for outcome 1
Measure: Number; unit: Encounters
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 108 | 121 | 308 | 290 | 420 | 417
Encounters
  Ambulance transport | 14 | 21 | 21 | 20 | 35 | 41
  Emergency room visits | 20 | 28 | 65 | 70 | 87 | 99
  Unscheduled outpatient visits | 513 | 579 | 1274 | 1216 | 1798 | 1834
  Home visits | 10 | 18 | 49 | 26 | 59 | 44
  Telephone calls | 51 | 76 | 112 | 117 | 163 | 196
  Advanced pulmonary function test | 16 | 20 | 35 | 26 | 51 | 46

15. Secondary Outcome: Asthma-related Healthcare Encounters by Type up to Week 52: Hospitalisations
Description: Broad-based healthcare utilisation asthma-related event information was collected by the Investigator/authorised delegate at each visit. At Visit 1, healthcare resource utilisation information was collected with a 1-year recall period; subsequent visits collected information with a recall period of 'since the last scheduled visit'. Total number of days spent in hospital was calculated across all patients for the following healthcare encounter category:
  • Hospitalisations (hospitalisations, intensive care and/or general care).
Time Frame: Baseline (Week 0) up to Week 52
Population: as for outcome 1
Measure: Number; unit: Days
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 108 | 121 | 308 | 290 | 420 | 417
Days | 82 | 175 | 334 | 414 | 417 | 590

16. Secondary Outcome: Asthma-related Healthcare Encounters by Type up to Week 52: Spirometry
Description: Broad-based healthcare utilisation asthma-related event information was collected by the Investigator/authorised delegate at each visit. At Visit 1, healthcare resource utilisation information was collected with a 1-year recall period; subsequent visits collected information with a recall period of 'since the last scheduled visit'. Total number of assessments was calculated across all patients for the following healthcare encounter category:
  • Spirometry.
Time Frame: Baseline (Week 0) up to Week 52
Population: as for outcome 1
Measure: Number; unit: Assessments
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Positive - Placebo | Biomarker Negative - Tralo 300 mg Q2W | Biomarker Negative - Placebo | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 108 | 121 | 308 | 290 | 420 | 417
Assessments | 148 | 151 | 284 | 270 | 434 | 426

17. Secondary Outcome: Serum Trough Concentration (Ctrough) of Tralokinumab During the Treatment Period up to Week 72
Description: To evaluate the pharmacokinetics (PK), pre-dose blood samples were collected at each visit and tralokinumab concentrations in serum were determined. Mean Ctrough concentrations are presented at each indicated visit up to Week 72.
Time Frame: Blood samples were collected pre-dose at Baseline (Week 0), and at Week 2, Week 8, Week 26, Week 56 (follow-up) and Week 72 (follow-up)
Population: All patients in the FAS who received tralokinumab and who had PK blood samples were included in the PK analysis set. Only patients in the biomarker positive and negative PK populations and with data available at the timepoints of testing were included in the analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/millilitre
Groups:
- Total - Tralo 300 mg Q2W: Tralokinumab 300 mg administered subcutaneously Q2W over a 52-week treatment period (up to 26 doses). 'Total' treatment arm represents all patients receiving tralokinumab in both the biomarker positive and biomarker negative patient populations.
Arm/Group | Biomarker Positive - Tralo 300 mg Q2W | Biomarker Negative - Tralo 300 mg Q2W | Total - Tralo 300 mg Q2W
Number analyzed (Participants) | 108 | 302 | 410
micrograms/millilitre
  Baseline | NA (NA) — Value was not calculable since below level of detection. | NA (NA) — Value was not calculable since below level of detection. | NA (NA) — Value was not calculable since below level of detection.
  Week 2: number analyzed (Participants) | 103 | 293 | 396
  Week 2 | 24.049 (172.475) | 20.916 (280.452) | 21.690 (248.876)
  Week 8: number analyzed (Participants) | 105 | 280 | 385
  Week 8 | 55.887 (206.478) | 52.324 (226.298) | 53.272 (220.301)
  Week 26: number analyzed (Participants) | 99 | 274 | 373
  Week 26 | 58.375 (145.256) | 47.707 (319.456) | 50.332 (264.686)
  Week 56 (follow-up): number analyzed (Participants) | 96 | 275 | 371
  Week 56 (follow-up) | 12.363 (591.282) | 12.513 (707.267) | 12.474 (671.922)
  Week 72 (follow-up): number analyzed (Participants) | 92 | 264 | 356
  Week 72 (follow-up) | 0.325 (251.436) | 0.384 (242.035) | 0.368 (244.398)

18. Secondary Outcome: Incidence Rate of Positive Anti-drug Antibodies (ADAs) Including the Characterization of Their Neutralizing Potential
Description: Assessments of ADA were performed using a tiered approach (screening, confirmatory and titering assays). Confirmed ADA positive samples were also tested for the presence of neutralising antibodies (nAb). ADA prevalence was defined as proportion of the study population having drug-reactive antibodies at any point in time. ADA incidence (treatment-emergent ADA) was defined as the sum of both treatment-induced (post-baseline ADA positive only) and treatment-boosted ADA. Persistently positive was defined as positive at ≥2 post-baseline assessments (with ≥16 weeks between first and last positive) or positive at last post-baseline assessment. Transiently positive was defined as having at least 1 post-baseline ADA positive assessment and not fulfilling the conditions of persistently positive. Treatment-boosted ADA was defined as baseline positive ADA titer that was boosted to a 4-fold or higher level following drug administration. Note: 'positive' is denoted by 'pos' in some category titles.
Time Frame: Baseline (Week 0), Week 26, Week 56 (follow-up) and Week 72 (follow-up)
Population: The ADA evaluable population included all patients in the safety analysis set (i.e. those who had received any IP) who had non-missing baseline ADA and at least 1 non-missing post-baseline ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 405 | 394
Participants
  ADA prevalence | 7 | 8
  ADA incidence | 5 | 3
  ADA positive at baseline | 2 | 5
  ADA positive post-baseline | 5 | 6
  ADA pos post-baseline and pos at baseline | 0 | 3
  ADA pos post-baseline and not detected at baseline | 5 | 3
  ADA not detected post-baseline and pos at baseline | 2 | 2
  Persistent Positive | 3 | 6
  Transient Positive | 2 | 0
  Treatment-boosted ADA | 0 | 0
  nAB positive at any visit | 5 | 2

ADVERSE EVENTS:
Time Frame: 72 weeks
Description: Serious and Other (non-serious) adverse event (AE) data is reported for the treatment period, from baseline (Week 0) to end of treatment (Week 52). Treatment-emergent AEs were defined with an onset date ≥ the first day of IP and ≤ (the last day of IP + 2 weeks). Patient population was the safety analysis set which included all patients who received at least one dose of IP.
  All-Cause mortality is reported for the overall study period (including the extended follow-up period), up to Week 72.
Arm/Group | Tralo 300 mg Q2W | Placebo
All-Cause Mortality (participants affected / at risk) | 1/425 | 4/422
Serious Adverse Events (participants affected / at risk) | 35/425 | 39/422
Other Adverse Events (participants affected / at risk) | 159/425 | 152/422
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tralo 300 mg Q2W (N=425) | Placebo (N=422)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis A (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis viral (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vascular headache (Nervous system disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Adnexa uteri pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 23 (30)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tralo 300 mg Q2W (N=425) | Placebo (N=422)
Injection site reaction (General disorders) | 23 (93) | 3 (5)
Bronchitis (Infections and infestations) | 34 (59) | 31 (50)
Upper respiratory tract infection (Infections and infestations) | 29 (49) | 31 (39)
Viral upper respiratory tract infection (Infections and infestations) | 50 (71) | 52 (80)
Headache (Nervous system disorders) | 40 (76) | 32 (49)
Asthma (Respiratory, thoracic and mediastinal disorders) | 35 (51) | 47 (79)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT02194699/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT02194699/SAP_001.pdf